## The Effect of Auricular Position on Measurement Values and Comfort in Measuring Body Temperature by Tympanic Way in Pediatric Patients

01.12.2022

## INFORMATION AND CONSENT DOCUMENT

You have been invited to participate in the research titled "The Effect of Auricular Position on Measurement Values and Comfort in Measuring Body Temperature by Tympanic Way in Pediatric Patients". This research was carried out by Hilal YILMAZ, a graduate of Istanbul University - Cerrahpasa Graduate Education Institute, Department of Fundamentals of Nursing, as a master's thesis, under the supervision of Assistant Professor Aylin ÖZAKGÜL. The aim of the study will be to determine the effect of placing the auricle position while measuring fever (body temperature) from the ear (tympanic route) on body temperature measurement values and comfort of patients in the measurements in pediatric patients aged 3-17 years. The patients we study will be randomly divided into two groups. Body temperature will be measured for one group without pulling the auricle first, then pulling it, and for the other group by pulling the auricle first and then without pulling. With an ear thermometer, your child's temperature will be measured without first pulling on the right ear, then pulling (positioning) or pulling the ear first and then without pulling. In addition, it will be asked whether he/she feels discomfort when the auricle is positioned, and if he/she does, how much he/she feels will be evaluated. In our study, our 19-question questionnaire will be applied to you, including your socio-demographic characteristics (age, occupation, educational status, etc.) and your knowledge about temperature measurement. Our research does not involve any risk.

Our research will take approximately 6 months. The estimated number of volunteers expected to participate in the study is 142.

Your child will be informed about this research in a way that he/she can understand and his/her consent will be obtained for participation in the research. It is entirely up to your free will to take part in this research, which has no side effects. Your decision not to participate will in no way adversely affect the health care and nursing care provided to you here. If you decide to participate, you can withdraw from the research at any time. This decision will not adversely affect the service provided.

The data we obtain will be used for scientific purposes and all information will be kept confidential. No payment will be made to you for your participation in this research, and you will not be charged any fees.

| 111 | hank | VOII |
|-----|-------|------|
| | Halik | vou |

Before starting the research above, I have read and understood the information given to me. I was also verbally informed about the research. Under these circumstances, I ACCEPT the invitation to participate in the research in question as a VOLUNTEER without any coercion or pressure.

A signed copy of this form will be given to me.

| Patient Relative's Name Surname: | Date: |
|----------------------------------|-------|
| Proximity: | |
| Signature: | |

## INFORMATION AND CONSENT DOCUMENT

Since you're in the hospital, the nurses will need to take your temperature. With a small thermometer in your right ear, we will take your temperature in just a few seconds. As we do this, we'll ask you how you're feeling. Can you let us to do this?

| Thank you very much. | |
|---|---|
| Hilal YILMAZ | |
| I have read and understood the information given to me above. I was also verbally ALLOW the nurse to take my temperature in my ear. A signed copy of this form will be given to me. | informed. I |
| Patient's name surname: Signature: | Date: |